CLINICAL TRIAL: NCT04357847
Title: Assessment of Endothelial and Haemostatic Changes During Severe SARS-CoV-2 Infection
Acronym: Covid-Thelium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, EBESNIER, Principal investigator, University Hospital, Rouen
Other Study IDs: 2020/097/OB
Record Dates: First submitted 2020-04-09; First posted 2020-04-22 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Covid-19; Endothelial Dysfunction; Thrombosis; Critically Ill
MeSH Terms: conditions — COVID-19; Thrombosis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The outbreak at covid-19 is caused by the SARS-CoV-2 virus. This virus can be responsible for severe respiratory failure but also for extra-respiratory organ dysfunctions associated with severe inflammatory stress. The endothelium is an important structure of the blood vessels and is implicated in the organ failure of many patients admitted in intensive care units. It could be affected by the virus and its alteration may explain the organ dysfunction of covid-19 ICU patients as well as the thrombotic processes frequently obstructed in this infection.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients admitted in ICU for covid-19 disease within the past 24 hrs

Exclusion Criteria:

* bactrial co-infection at admission
* expected death within the next 24 hrs
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with documented SARS-CoV-2 infection (PCR or CTscan)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Association of InterCellular Adhesion Molecule-1 plasma level with 28 days mortality | 24 hours
  Plasma of covid-19 patients will be tested for endothelial injuries, notably with the measurement of InterCellular Adhesion Molecule 1 level by Enzym-Linked Immunosorbent Assay. The association of these levels with 28-days mortality will be evaluated as prognosis markers.

SECONDARY OUTCOMES:
Association of Endothelin-1 plasma level with 28 days mortality | 24 hours
  Endothelin-1 will be assessed in blood as a maker of endothelial injuries, expressed in pg/mL. its association with 28 -days mortality will be evaluated.
Association of Vascular Endothelial Growth Factor A plasma level with 28 days mortality | 24 hours
  Vascular Endothelial Growth Factor A plasma level will be measured in blood as a marker of endothelial injury expressed in pg/mL. its association with 28 -days mortality will be evaluated.
Association of soluble Vascular Endothelial Growth Factor Receptor type 1 with 28 days mortality | 24 hours
  This soluble receptor is another marker of endothelial injury and will be measured in blood and expressed as pg/mL. Its association with 28-days mortality will be evaluated.
Association of syndecan -1 plasma level with 28 days mortality | 24 hours
  syndecan -1 is a marker of degradation of glycocalyx, raised during endothelial injury. It will be measured in blood and expressed as pg/mL. Its assocation with 28-days mortality will be evaluated.
Association of D-dimers plasma levels with thrombotic events | 24 hours
  D-dimers si marker of enhanced thrombotic activity. It may be increased during covid-19 disease but its correlation with endothelial injury is not known. It will be measured in blood and expressed as microgrammes/L, and then correlated with ICAM-1 plasma levels
Association of von Willebrandt Factor with thrombotic events | 24 hours
  This marker may be raised during endothelial injury and may explained thrombotic status of covid-19 patients. Its blood levels will be measured and expressed as international unit/dL, and correlated with ICAM-1 plasma levels
Association of Viscoelastic testing with thrombotic events | 24 hours
  Clot Stiffness and its fibrinogen and platelet contributions (expressed in kPa) will be measured as novative approach, using Quantra (Stago Inc) device, to explore hemostasis alterations of covid-19 patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided